CLINICAL TRIAL: NCT04061122
Title: The Role of Congenital Mucosal Immune System in the Airways of Patients With COPD
Brief Title: The Role of Congenital Mucosal Immune System in the Airways of Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Pawel Majak, Principal Investigator, Medical University of Lodz
Other Study IDs: RNN/206/16IKE
Record Dates: First submitted 2019-08-12; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: COPD Exacerbation; Smoking, Tobacco
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- EX + / ECTS +: Patients suffering COPD exacerbation in last 7 days; active tobacco smokers
  Interventions: Diagnostic Test: airway epithelial smear test
- EX - / ECTS +: Patients without COPD exacerbation in last 6 months; active tobacco smokers
  Interventions: Diagnostic Test: airway epithelial smear test
- EX + / ECTS -: Patients suffering COPD exacerbation in last 7 days; quited tobacco smoking at least 12 months earlier
  Interventions: Diagnostic Test: airway epithelial smear test
- EX - / ECTS -: Patients without COPD exacerbation in last 6 months; quited tobacco smoking at least 12 months earlier
  Interventions: Diagnostic Test: airway epithelial smear test

INTERVENTIONS:
Diagnostic Test: airway epithelial smear test — all patients will be subjected to all scheduled procedures: airways epithelial smear test, measurement of VOCs in exhaled air and airways slide sample culture
  Other Names: measurement of VOCs; culture

SUMMARY:
The purpose of the study is to explore the role of congenital mucosal immune system in the airways of patients with COPD including the impact of ILCs (Innate lymphoid cells) on metabolism of epithelial cells.During the research the following methods will be applied: measurement of Volatile Organic Compounds (VOCS), airway epithelial cytology and culture.

DETAILED DESCRIPTION:
ILCs profiles, epithelium metabolism measured by VOCS and microbiome profiling (specific 16S rRNA-16S ribosomal RNA gene-targeted qPCR) will by determined in the airways of patients with COPD after the exacerbation. Microbiome profiling will be based on next generation sequencing (NGS) of the 16S rRNA encoding region.

ELIGIBILITY:
Exclusion Criteria:

* Neoplasm
* Diabetes
* Astma
* acute airway infection in last 2 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EX (COPD exacerbation) TS (tobacco smoking)
  Group: EX + / TS + Patients suffering COPD exacerbation in last 7 days; active tobacco smokers
  Group: EX - / TS + Patients without COPD exacerbation in last 6 months; active tobacco smokers
  Group: EX + / TS - Patients suffering COPD exacerbation in last 7 days; smoking was stopped a minimum of 12 months before the first visit
  Group: EX - / TS - Patients without COPD exacerbation in last 6 months; smoking was stopped a minimum of 12 months before the first visit
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
percentage of nasal ILCs (Innate lymphoid cells) after COPD exacerbation | through study completion, an average of 1 year
  The assessment of the nasal mucosa material after COPD exacerbation will include: percentage of ILC1, 2 and 3 cells (immunophenotyping and measurement by flow cytometry)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Asthma and Allergy, Barlicki University Hospital, Medical University of Lodz, Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No